CLINICAL TRIAL: NCT04246099
Title: Effect of Opioid-free Anesthesia on Perioperative Period After Video-assisted Thoracoscopic Lobectomy: a Retrospective Study
Brief Title: Opioid-free Anesthesia in Thoracic Surgery
Acronym: VATOFA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: VATOFA
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Thoracic; Surgery
Keywords: Post-operative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group opioid free anesthesia: Patient benefit of the opioid free anesthesia protocol
  Interventions: Other: Post-operative care
- Group opioid based anesthesia: Patient don't benefit of the opioid free anesthesia protocol
  Interventions: Other: Post-operative care

INTERVENTIONS:
Other: Post-operative care — Retrospective collection of clinical data recorded in the electronic medical record.
  The following variables were continuously recorded in the institutional database: age, gender, body weight, height, personal medical history, American Society of Anesthesiologists (ASA) score, type of thoracic surgery, the duration of surgery, duration of anesthesia (from intubation to extubation), the duration of PACU stay, the need for morphine titration, epinephrine, norepinephrine.
  For data at day 30, the vast majority of patients were included in the enhanced recovery program and as such benefited from a consultation at 1 month with a coordination nurse who collected data on post-operative pain in a standardized manner.
  All data was extracted from investigators institutional database and collected by a physician who was not involved in the care of the study patients.

SUMMARY:
No study has been conducted to demonstrate the feasibility and safety of an Opioid-Free Anesthesia (OFA) protocol compared to Opioid-Based Anesthesia (OBA) in thoracic surgery, at risk for intense post-operative pain, to improve patient care. The aim of the present study was to evaluate the effect of OFA on post-operative opioids consumption, pain and the post-operative period after lobectomy by Video-Assisted Thoracoscopy Surgery (VATS). systems.

Investigators perform a retrospective, single-center study in 2019. Patients were divided into two groups: OFA (with dexmedetomidine) or OBA (sufentanyl).

Investigators analyse the total postoperative opioid consumption in the 48 h after surgery. Investigators asses pain intensity in the 48 h after surgery, operative hemodynamic stability, Post-Operative Pain (POP) in Post-Anesthesia Care Unit (PACU) and POP on day 30.

All data are available in the medical record

Hypothesis: OFA can reduce post-operative opioids consumption, pain in lobectomy by video-assisted thoracoscopy surgery (VATS).

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients admitted for lobectomy or wedge video-assisted thoracoscopy
* Opioid Free Anesthesia (OFA) administration was left to the discretion of the attending anesthetist according to his or her practices and habits.
* age 18 or over
* lobectomy or wedge resection by Video-Assisted Thoracoscopy Surgery (VATS)

Exclusion Criteria:

* toxicomania,
* epidural analgesia use,
* thoracotomy conversion
* Patient-Controlled Analgesia with morphine (PCA)
* Patient who object to take part of the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All consecutive patients admitted for lobectomy or wedge video-assisted thoracoscopy in Department of Anesthesiology and Intensive Care at Louis Pradel University Hospital.
  If patient benefit of the OFA protocol, he was part of the group OFA (opioid free anesthesia) If patient don't benefit of the OFA protocol, he was part of the group OBA (opioid based anesthesia)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Cumulative dose of postoperative opioid | 48 hours
  The primary endpoint was the cumulative dose of postoperative opioid in the first 48 h (D2) (in milligrams of oral morphine equivalent) which included morphine and tramadol after conversion (1mg of intra-veinous morphine = 3 mg of oral morphine, and 10 mg of oral morphine = 50 mg of oral tramadol)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Intensive Care - Louis Pradel University Hospital - Hospices Civils, Lyon, France, Bron, France

IPD SHARING:
Plan to Share IPD: No